CLINICAL TRIAL: NCT05271773
Title: Impact of Therapeutic Intervention on Quality of Life in Patients With Ulcerative Colitis Depending on the Mucosal Healing Degree
Brief Title: Impact of Therapeutic Intervention on Quality of Life in Patients With Ulcerative Colitis
Acronym: CAVI_CU
Status: Completed | Type: Observational
Sponsor: Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (Other)
Responsible Party: Sponsor
Other Study IDs: CAVI_CU
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: IBD-Inflammatory Bowel Disease; UC - Ulcerative Colitis
Keywords: PRO- patient reported outcomes; HRQOL - health-related quality of life; mucosal healing; ASA - acetylsalicylic acid; CRP - C reactive protein; IBDQ - Inflammatory Bowel Disease Questionnaire; SPSS
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stool specimen (Fecal calprotectin)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mayo 0: Patients with an established diagnosis of UC through regular criteria (clinical, analytical, endoscopic, radiological and/or histological ones), in clinical remission (partial Mayo score ≤2) for at least three months, who had undergone surveillance colonoscopy after 12 months from the study outset, with a Mayo 0 endoscopic activity.
- Mayo 1: Patients with an established diagnosis of UC through regular criteria (clinical, analytical, endoscopic, radiological and/or histological ones), in clinical remission (partial Mayo score ≤2) for at least three months, who had undergone surveillance colonoscopy after 12 months from the study outset, with a Mayo 1 endoscopic activity.

SUMMARY:
This study is therefore postulated as a clear alternative that evaluates patients´quality of life, and recognises fecal calprotectin as an inflammatory marker.

Longitudinal, prospective, multi-center cohort study to measure the impact that the therapeutic attitude (treatment intensification/de-intensification o escalation/de-escalation) has on the quality of life of patients with UC given a colonoscopy revealing mucosal healing (Mayo 0, Mayo 1); considering as treatment intensification/de-intensification a dose increase or decrease on the same line of treatment, and escalation/de-escalation if there is a change to a new line of treatment.

DETAILED DESCRIPTION:
Research justification: There is not enough evidence on the effect of therapeutic intervention implemented by doctors in patients with IBD, depending on the rate of mucosal healing at colonoscopy.

From previous studies the investigators know that patients with a Mayo 1 endoscopic score are at a much greater risk for developing a disease outbreak, thus requiring a treatment escalation more frequently than those Mayo 0 patients. Then, it is needed a study of real clinical practice to evaluate the efficacy of this therapeutic intervention (same treatment or escalation/de-escalation strategy) in patients' quality of life.

Objectives:

Primary:

- After 6 and 12 months, to measure the impact that the therapeutic attitude (treatment intensification/de-intensification o escalation/de-escalation) has on the quality of life of patients with UC given a colonoscopy revealing mucosal healing (Mayo 0, Mayo 1); considering as treatment intensification/de-intensification a dose increase or decrease on the same line of treatment, and escalation/de-escalation if there is a change to a new line of treatment.

Secondary:

* To evaluate the impact of inflammatory markers at the end of 6 and 12 months (C-reactive protein, fecal calprotectin).
* Outbreak risk assessment depending on the intervention developed (same treatment, or escalation/de-escalation).

Study design: Longitudinal, prospective, multi-center cohort study. Target population. Patients with an established diagnosis of UC through regular criteria (clinical, analytical, endoscopic, radiological, and/or histological ones), in clinical remission (partial Mayo score ≤2) for at least three months, who had undergone surveillance colonoscopy after 12 months from the study outset, with a Mayo 0 or Mayo 1 endoscopic activity.

The coverage of the data collections shall extend to all centers via the REDCap platform. The basal characteristics studied are date of birth and gender, and data associated with characteristics of UC such as date of diagnosis, the extent of the area affected, and ongoing treatment when the assessment is performed (5-ASA, immunomodulatory, and/or biologics).

A short 9-item version of the IBD Questionnaire together with an IBD-Control one will be used to register changes across the treatment course at the moment of inclusion (basal), for a maximum period of 2 weeks after colonoscopy. CRP and fecal calprotectin values (both analyzed by each center considering quantitative data) shall be calculated in proportion to the period from 2 weeks prior and 2 weeks after colonoscopy (preventing from collecting feces samples during colonoscopy preparation).

Physicians will schedule follow-up appointments to obtain both an IBDQ-9 and an IBD-Control questionnaire and to monitor CRP and fecal calprotectin values as well as changes in treatment at that moment; to identify the appearance in that period of any clinical outbreak (defined as the presence of rectal bleeding together with any of these: need of any remission-induction therapy -including topical treatment-, any treatment escalation -increasing dose levels, topical medication included, or any change in treatment- and requiring hospitalization or colectomy).

Sample size planning: At the 95% confidence level and a power of 80%, with a one-sided hypothesis:

* To demonstrate a difference in recurrence with no treatment changes, by assuming a recurrence of 36.6% from the Mayo 1 group, and of 9.4% from Mayo 0 group (8), the investigators need 28 patients in each group.
* To demonstrate that due to increased treatment, Mayo 0 group does not get better and Mayo 1 group will show a 25% of improvement compared to the no changes-in-treatment plan, a sample of 57 patients per group is needed.
* To demonstrate that treatment reduction increases recurrence up to 10% in Mayo 0 group of patients and to 40% in Mayo 1 group compared to the no changes-in-treatment plan, a sample of 14 patients per group is needed.

Statistical methods. An electronic anonymized database will save the codified data obtained. Demographic and clinical variables will be characterized by descriptive statistics parameters. Quantitative variables will be measured by medians and interquartile ranges or means and standard deviation. Qualitative variables will take into account absolute and relative frequencies (%), and 95% confidence interval. Statistical tests will be performed using STATA 15 and IBM SPSS Statistics 25 statistical software packages.

ELIGIBILITY:
Inclusion Criteria:

* UC diagnosed.
* Age ≥ 18.
* Signed and dated informed consent form.
* Have undergone a Mayo 0 or 1 endoscopic score colonoscopy while in clinical remission.

Exclusion Criteria:

* Incomplete colonoscopy.
* Previous bowel resection.
* Ostomy patient.
* Active infection.
* Pregnancy.
* Lack of patient's informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an established diagnosis of UC through regular criteria (clinical, analytical, endoscopic, radiological and/or histological ones), in clinical remission (partial Mayo score ≤2) for at least three months, who had undergone surveillance colonoscopy after 12 months from the study outset, with a Mayo 0 or Mayo 1 endoscopic activity.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
To measure the impact that the therapeutic attitude, based on IBDQ9 and IBD control questionaire, has on the quality of life of patients with UC given a colonoscopy revealing mucosal healing | at 6 and 12 months
  After 6 and 12 months, to measure the impact that the therapeutic attitude (treatment intensification/de-intensification o escalation/de-escalation) has on the quality of life of patients with UC given a colonoscopy revealing mucosal healing (Mayo 0, Mayo 1); considering as treatment intensification/de-intensification a dose increase or decrease on the same line of treatment, and escalation/de-escalation if there is a change to a new line of treatment.

SECONDARY OUTCOMES:
To evaluate the impact of inflammatory markers | at 6 and 12 months
  To evaluate the impact of inflammatory markers at the end of 6 and 12 months (C-reactive protein, fecal calprotectin).
Outbreak risk assessment depending on the intervention developed | at 6 and 12 months
  Outbreak risk assessment depending on the intervention developed (same treatment, or escalation/de-escalation).

CONTACTS AND LOCATIONS:
Overall Officials: GETECCU GETECCU, Study Chair — Grupo Español de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa
Locations (10):
- Spain (10):
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitari Parc Taulí, Sabadell, Catalonia
  - Hospital de Santa Bárbara de Puertollano, Puertollano, Ciudad Real
  - Hospital Universitario de Cáceres, Cáceres, Extremadura
  - Hospital Universitario de Santiago de Compostela, Santiago de Compostela, Galicia
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario. Miguel Servet, Zaragoza